CLINICAL TRIAL: NCT06137950
Title: Interferon Alpha Therapy for Cervical CIN I and HPV Infection
Brief Title: Interferon Alpha Therapy for Cervical CINI and HPV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mongolian National University of Medical Sciences (Other)
Collaborators: Mongolian National Cancer Center (Unknown)
Responsible Party: Principal Investigator, Batsuren Choijamts, Head of department, Mongolian National University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNUMS2021100701
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cervical Dysplasia; HPV Infection
Keywords: CIN I, HPV infection
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections | interventions — Interferon alpha-2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Interferon α2b gel treatment for 30 days.
  Interventions: Drug: gel Interferon arm
- Treatment (Experimental): Interferon α2b gel treatment for 30 days
  + Interferon α2b 3 MIU rectal suppository for 10 days
  Interventions: Drug: gel Interferon arm; Drug: gel Interferon and interferon suppository arm

INTERVENTIONS:
Drug: gel Interferon arm — 0.2 ml gel interferon will be administered into vaginal using 1 ml syringe with measurement line. Patients will be trained how to fill the syringe and put into the vagina. Gel will be administered 2 times per day during the non menstruating day totally for 28 days.
  Other Names: Interferon alfa-2b low dose local treatment
Drug: gel Interferon and interferon suppository arm — 0.2 ml gel interferon will be administered into vaginal using 1 ml syringe with measurement line. Patients will be trained how to fill the syringe and put into the vagina. Gel will be administered 2 times per day during the non menstruating day totally for 28 days.
  3MIU suppository will be given to patients and will be trained how to use. Each patient in the arm will use the suppository twice a day for 10 days with vaginal therapy.
  Other Names: Interferon alfa-2b low dose local and high dose systemic treatment
  Arms: Treatment

SUMMARY:
Mongolia is a traditionally nomadic and population is scarce in rural areas. Thus, the medical care service is not sufficient. In 2000, Mongolian government has developed and implemented the millennium project in cooperation with WHO. During the years pap smear analysis of implemented in all rural areas and clinicians, lab technicians have been taught for the cervical cancer screening. However, the project has finished in 2015 and the rural and district hospitals has lost the trained professionals. Still the cervical cancer is in second place after liver cancer in women.

The purpose of the study is to identify the type of HPV genotype and to treat the HPV infection by local interferon α2b.

Materials and methods: HPV positive patients will be enrolled to the study. HPV genotype will be determined by the PCR in laboratory. Pap smear will be taken and staged by the CIN. Pathological tissue will be taken under colposcopy with acetic acid test. Follow up visit will be done on 10th, 30th days of the treatment.

At the end of 90th days of treatment, pap and histology test will be repeated and CIN regression or viral eradication will be evaluated.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy of interferon treatment for HPV infection shedding and early CIN change.

Women aging from 20-40 years will be enrolled in the study. The treatment will be held in two arms. One arm will be administered only vaginal gel interferon treatment. The other arm will receive both vaginal gel interferon and rectal suppositories with interferon dosing 3,000,000 IU.

In the beginning of the study all patient will have cervical pap smear and HPV typing.

HPV testing will be done using real time PCR method to determine the subtype of HPV (16,18,31,33,35,39,45,51,52,56,59,68).

At the beginning and at the end of the study all patient will have histology test.

Histology test will be done Giemsa staining and evaluated by WHO 2014 classification of cervical histology including CINI, CINII, CINIII, cervical cancer in situ and further.

Pap smear will be evaluated by Bethesda classification. Immunohistology staining will be done on the cervical tissue using anti-CD3 and anti-CD19 to evaluate the B cell invasion into the cervix.

ELIGIBILITY:
Inclusion Criteria:

* Pap smear LSIL
* HPV infection positive
* No anti-viral treatment in 2 weeks before treatment

Exclusion Criteria:

* No consent has obtained
* Anti-viral treatment in 2 weeks
* Breastfeeding or pregnant

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is about treatment of uterine cervical dysplasia
Enrollment: 60 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Pap smear | 90 days
  LSIL, HSIL or regression of the change will be assessed.
Colposcopic change | 90 days
  Cervical changes before and after treatment will be compared.

SECONDARY OUTCOMES:
Histopathologic change | 90 days
  CINI, CINII or regression of the cervical dysplasia will be evaluated.
Immunohistochemical change | 90 days
  Anti CD-3 and anti CD-19 staining will be done and stained cells will be calculated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Batsuren Choijamts, Ph.D, Principal Investigator — Mongolian National University of Medical Science
Locations (1):
- National Cancer Center, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nestor MS, Gold MH, Kauvar AN, Taub AF, Geronemus RG, Ritvo EC, Goldman MP, Gilbert DJ, Richey DF, Alster TS, Anderson RR, Bank DE, Carruthers A, Carruthers J, Goldberg DJ, Hanke CW, Lowe NJ, Pariser DM, Rigel DS, Robins P, Spencer JM, Zelickson BD. The use of photodynamic therapy in dermatology: results of a consensus conference. J Drugs Dermatol. 2006 Feb;5(2):140-54. PMID 16485882
- [Background] Hoffman SR, Le T, Lockhart A, Sanusi A, Dal Santo L, Davis M, McKinney DA, Brown M, Poole C, Willame C, Smith JS. Patterns of persistent HPV infection after treatment for cervical intraepithelial neoplasia (CIN): A systematic review. Int J Cancer. 2017 Jul 1;141(1):8-23. doi: 10.1002/ijc.30623. Epub 2017 Feb 27. PMID 28124442
- [Background] Shi HJ, Song H, Zhao QY, Tao CX, Liu M, Zhu QQ. Efficacy and safety of combined high-dose interferon and red light therapy for the treatment of human papillomavirus and associated vaginitis and cervicitis: A prospective and randomized clinical study. Medicine (Baltimore). 2018 Sep;97(37):e12398. doi: 10.1097/MD.0000000000012398. PMID 30213012
- [Background] Su Y, Zhang M, Zhang W, Shi H. Clinical efficacy of cryotherapy combined with interferon in the treatment of chronic cervicitis complicated with HPV infection. Pak J Pharm Sci. 2017 Jul;30(4(Suppl.)):1505-1508. PMID 29044006